CLINICAL TRIAL: NCT05915208
Title: Histiocytic Disorder Follow-up Study
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gaurav Goyal, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300008744
Record Dates: First submitted 2023-05-25; First posted 2023-06-22 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Histiocytosis; Langerhans Cell Histiocytosis; Erdheim-Chester Disease; Rosai Dorfman Disease; Xanthogranuloma; Malignant Histiocytoses
Keywords: survivorship; long-term; targeted therapy; second cancer
MeSH Terms: conditions — Histiocytosis; Histiocytosis, Langerhans-Cell; Erdheim-Chester Disease; Histiocytosis, Sinus; Histiocytic Sarcoma; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of the study is to describe the burden of chronic health conditions, psychological dysfunction, chronic pain, healthcare utilization, worse health-related quality of life, overall mortality, and cause-specific mortality among individuals with histiocytic disorders

DETAILED DESCRIPTION:
Background

Over the last decade, major advances have occurred in histiocytic disorders with the discovery of MAPK-ERK pathway mutations leading to targeted therapeutics using BRAF- and MEK-inhibitors. However, there is a lack of large studies informing the burden of morbidity and mortality among people with histiocytosis. Institutional studies in pediatric LCH suggest that survivors suffer from long-term impairment of health related quality of life, cognitive dysfunction, pituitary dysfunction, and hearing difficulties in 20-50% cases. Studies from the investigative team and others have also shown a high incidence of acute myeloid leukemia and other second primary malignancies in pediatric and adult LCH. Chronic medical conditions may arise as a function of the disease biology or due to cancer therapy, as seen in other hematologic malignancies.

Design

Retrospective cohort study aimed at determining the risk of chronic health conditions and cause-specific mortality in pediatric and adult patients with histiocytic disorders. The study will include patients from the Histiocytosis Association registry and other institutions including UAB (n~6000). The participants will complete a validated questionnaire capturing details of chronic health conditions, health related quality of life, cognitive/psychological function, and healthcare utilization.

Future directions

The results from our study will be instrumental in formulating follow-up guidelines for histiocytic disorders and developing targeted survivorship programs to improve overall outcomes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of histiocytic disorder at any age

  1. Langerhans cell histiocytosis,
  2. Erdheim-Chester disease,
  3. Rosai-Dorfman disease,
  4. Xanthogranuloma,
  5. Mixed histiocytosis
  6. Malignant histiocytosis (Histiocytic sarcoma, langerhans cell sarcoma, interdigitating cell sarcoma)
  7. Hemophagocytic lymphohistiocytosis

Exclusion Criteria:

* None

Ages: 0 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with diagnosis of histiocytic disorder are eligible to participate, including family members (next of kin) of deceased individuals.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Chronic health conditions diagnosed after LCH diagnosis graded using the Common Terminology Criteria for Adverse Events (CTCAE), v5.0 (https://ctep.cancer.gov) | From diagnosis of histiocytic disorder to age at completion of survey, assessed up to 200 months
  The CTCAE criteria for CHCs distinguishes each acute and chronic condition (including SPMs) in persons with cancer from grades 1 through 4 with unique clinical descriptions of severity (grade 1, mild; grade 2, moderate; grade 3, severe; grade 4, life-threatening/disabling). The main outcome will be the number of distinct CTCAE grade 3-4 conditions among LCH cases compared with unaffected (non-cancer) controls.
All-cause and cause-specific mortality | 2 years preceding death
  Causes of death will be grouped into primary cancer (LCH)-related mortality (PCRM) and non-primary cancer-related mortality (NPCRM - death from all causes other than the index LCH diagnosis) by two independent investigators.

SECONDARY OUTCOMES:
Factors associated with new-onset morbidity | From diagnosis to age at completion of survey, assessed up to 200 months
  We will build a prediction model that has a good discrimination for predicting CHC, SPMs, and psychological outcomes separately using data from the LCH (case) cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Goyal, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided